CLINICAL TRIAL: NCT01670487
Title: Prospective,Randomized,Blinded, Comparative,Efficacy and Safety Trial of Vapocoolant (Pain Ease Medium Stream) for Intravenous Cannulation in Emergency Department Patients.
Brief Title: Vapocoolant (Pain Ease Medium Stream) for Intravenous Lines in Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Gebauer Company (Network)
Responsible Party: Principal Investigator, Sharon Mace, Staff Physician & Research Director, Emergency Services Institute, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GEB-02
Record Dates: First submitted 2012-08-13; First posted 2012-08-22 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: Vapocoolant
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vapocoolant (Pain Ease Medium Stream) (Active Comparator): Application of the stream steadily 4 to 10 seconds onto the cannulation site.
- Nature's Tears (Placebo Comparator): Apply sterile water (see manufacturer above) steadily 4-10 seconds onto the cannulation site.
  Interventions: Device: Sterile water

INTERVENTIONS:
Device: Vapocoolant — Topical stream of 4 to 10 seconds duration to skin
  Other Names: Pain Ease stream
Device: Sterile water — Topical intervention of sterile water stream 4 to 10 seconds to skin.
  Other Names: Nature's Tears by Bio-Logic Aqua Technologies
  Arms: Nature's Tears

SUMMARY:
To determine the efficacy and safety of vapocoolant stream (Pain Ease Medium Stream ) in decreasing the pain of intravenous cannulation.

To compare vapocoolant stream (Pain Ease medium Stream) with control (e.g. sterile water) stream.

DETAILED DESCRIPTION:
Vapocoolant sprays have been used to decrease the pain associated with painful medical procedures such as immunizations, needle aspirations, injections, venipuncture and intravenous cannulation. In general, vapocoolant sprays , have been found to be effective in decreasing the pain of various medical procedures. Moreover, the use of vapocoolant sprays ,unlike other local anesthetics , such as infiltrative lidocaine , is not associated with a painful injection and does affect the success rate of the procedure including intravenous cannulation and may even increase the success rate of the intravenous cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing intravenous cannulation
* Adults age 18 years equal or greater than.
* Stable patient
* Mentally competent patient able to understand the consent form

Exclusion Criteria:

* Patients with any allergies to the spray components ( e.g.1,1,3,3, pentafluoropropane or 1,1,1,2 tetrafluoroethane )
* Critically ill or unstable patient (e.g. sepsis or shock)
* Infants and children of age , <18 years.
* Pregnant
* Intravenous cannulation site located in area of compromised blood supply. (ex: patients with Peripheral Vascular Disease , Raynaud's disease, gangrene, Buerger's disease)
* Intravenous cannulation site located in area of insensitive skin; such as , patients with a peripheral neuropathy including diabetic neuropathy.
* Patient intolerant of cold or with hypersensitivity to the cold.
* Patient unable or unwilling to give consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon E. Mace, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hijazi R, Taylor D, Richardson J. Effect of topical alkane vapocoolant spray on pain with intravenous cannulation in patients in emergency departments: randomised double blind placebo controlled trial. BMJ. 2009 Feb 10;338:b215. doi: 10.1136/bmj.b215. PMID 19208703
- [Background] Page DE, Taylor DM. Vapocoolant spray vs subcutaneous lidocaine injection for reducing the pain of intravenous cannulation: a randomized, controlled, clinical trial. Br J Anaesth. 2010 Oct;105(4):519-25. doi: 10.1093/bja/aeq198. Epub 2010 Aug 3. PMID 20682573
- [Background] Biro P, Meier T, Cummins AS. Comparison of topical anaesthesia methods for venous cannulation in adults. Eur J Pain. 1997;1(1):37-42. doi: 10.1016/s1090-3801(97)90051-3. PMID 15102427
- [Background] Hartstein BH, Barry JD. Mitigation of pain during intravenous catheter placement using a topical skin coolant in the emergency department. Emerg Med J. 2008 May;25(5):257-61. doi: 10.1136/emj.2006.044776. PMID 18434455
- [Background] Baxter AL, Leong T, Mathew B. External thermomechanical stimulation versus vapocoolant for adult venipuncture pain: pilot data on a novel device. Clin J Pain. 2009 Oct;25(8):705-10. doi: 10.1097/AJP.0b013e3181af1236. PMID 19920721
- [Background] Patterson P, Hussa AA, Fedele KA, Vegh GL, Hackman CM. Comparison of 4 analgesic agents for venipuncture. AANA J. 2000 Feb;68(1):43-51. PMID 10876451
- [Derived] Barbour T, O'Keefe S, Mace SE. Topical Refrigerant Spray for IVs: Patient/Provider Responses - Prospective, Double-blind, Randomized Study. West J Nurs Res. 2021 Aug;43(8):762-769. doi: 10.1177/0193945920976061. Epub 2020 Dec 8. PMID 33292081
- [Derived] Mace SE. Prospective, double blind, randomized, controlled trial comparing vapocoolant spray versus placebo spray in adults undergoing intravenous cannulation. Scand J Pain. 2017 Oct;17:8-15. doi: 10.1016/j.sjpain.2017.06.002. Epub 2017 Jul 10. PMID 28850378

RESULTS

PARTICIPANT FLOW:
Groups:
- Vapocoolant (Pain Ease Medium Stream): Application of the stream steadily 4 to 10 seconds onto the cannulation site.
  Vapocoolant: Topical stream of 4 to 10 seconds duration to skin
Period: Overall Study
Arm/Group | Vapocoolant (Pain Ease Medium Stream) | Nature's Tears
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: adults undergoing IV annulation in ED
Groups:
- Vapocoolant (Pain Ease Medium Stream): Applied Vapoccolant in a topical stream of 4 to 10 seconds duration to skin
- Nature's Tears: Applied Nature's Tears in a topical stream of 4 to 10 seconds duration to skin
- Total: Total of all reporting groups
Arm/Group | Vapocoolant (Pain Ease Medium Stream) | Nature's Tears | Total
Number analyzed (Participants) | 150 | 150 | 600
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  number analyzed (Participants) | 150 | 150 | 300
  (all) | 52 [35 to 60] | 50 [37 to 62] | 51 [35 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 150 | 150 | 300
  Female | 94 | 64 | 158
  Male | 56 | 86 | 142

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on the Numeric Rating Scale (NRS)
Description: Numeric rating scale (NRS) 0-10 : 0 (no pain) - 5 (moderate pain) - 10 (worst pain). Scores to be utilized after stream device applied and after intravenous catheter placement.
Time Frame: pain of intravenous catheter placement.
Population: adults undergoing placement of an intravenous line in the emergency department
Measure: Mean (Standard Deviation); unit: NRS
Groups:
- Placebo (Nature's Tears): Application of the stream steadily for 4 to 10 seconds
Arm/Group | Vapocoolant (Pain Ease Medium Stream) | Placebo (Nature's Tears)
Number analyzed (Participants) | 150 | 150
NRS | 2.3 (2.4) | 4.3 (3.0)

ADVERSE EVENTS:
Arm/Group | Vapocoolant (Pain Ease Medium Stream) | Nature's Tears
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 16/150 | 2/150
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vapocoolant (Pain Ease Medium Stream) (N=150) | Nature's Tears (N=150)
skin irritation such as redness or blanching (Skin and subcutaneous tissue disorders) | 16 (16) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No